CLINICAL TRIAL: NCT06706453
Title: Sleep Survey for Medical Trainees: a Collaboration Between the World Sleep Society and National Sleep Centre / Sleep Societies
Brief Title: Sleep Survey for Medical Trainees
Acronym: SSMT
Status: Enrolling by invitation | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: MRA-23/24-45277
Record Dates: First submitted 2024-09-11; First posted 2024-11-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Sleep; Shift Work; Circadian Rhythm; Sleep Apnea; Insomnia
Keywords: Medical training; on call; working time
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Medical staff: Anyone who works in medicine with any on call commitment (student, intern, fellow, resident, consultant)

SUMMARY:
Background

This is a survey to understand sleep in the context of medical trainees (on call) and the participants knowledge about the relevance of sleep, shiftwork, and the impact that sleep may have on their working performance. The survey has been developed by sleep experts from America, Europe, and Africa, in collaboration with the World Sleep Society. It should take about 30-40 minutes to complete.

The survey will focus on three different aspects, complemented by two standard questionnaires:

1. Demographics and Place of Work
2. Basic Knowledge and Perception of Sleep
3. Sleep Routine
4. Epworth Sleepiness Scale, Insomnia Sleep Inventory

ELIGIBILITY:
Inclusion Criteria:

* medical staff
* student / intern / fellow / resident / consultant
* delivering on call work
* any gender

Exclusion Criteria:

* non-medical staff working in hospitals from the wider multidisciplinary team
* underage (less than 18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical staff that undertakes on call work (medical student, intern, fellow, resident, consultant)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Impact of being ON CALL in the hospital on sleep | cross-sectional survey (while filling in the questionnaire); experience within 3 months of completion
  Composite outcome as described by deviation from regular sleep in terms of sleep quality (points, out of 10; higher scores indicating more symptoms), quantity (duration, hours:mins), and deviation from circadian rhythm (measured in times of the day and duration, as well as perceived disturbance, points out of 10; higher points indicating more symptoms)

SECONDARY OUTCOMES:
Demographics | within 3 months of completion of survey
  Basic demographics, family status/children
Sleep routine | within 3 months of completion of survey
  Sleep routine while ON CALL / not ON CALL (bed time, hours:mins; wake up time, hours:mins)
Epworth Sleepiness Scale | within 3 months of completion
  Validated screening questionnaire containing eight questions related to likelihood of dozing (min score 0, max score 24 points; higher scores indicate more symptoms)
Insomnia Severity Index | within 3 months of completion
  Validated questionnaire assessing likelihood of insomnia (7 questions, min 0 / max 28 points; higher scores indicate more symptoms)
Basic knowledge and perception of sleep | within 3 months of completion of survey
  Impact of work/on call on sleep (duration of sleep, hours:mins; sleep quality, points out of 10; symptoms, points out of 10; higher scores indicating more symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Kings College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Acquired data may be subject to underlying legislation (according to country, e.g. GDPR). In reasonable cases and upon written request / following ethics committee approval data sharing for the purpose of IPD analysis will be considered case-by-case.

REFERENCES:
- [Background] Lim DC, Najafi A, Afifi L, Bassetti C, Buysse DJ, Han F, Hogl B, Melaku YA, Morin CM, Pack AI, Poyares D, Somers VK, Eastwood PR, Zee PC, Jackson CL; World Sleep Society Global Sleep Health Taskforce. The need to promote sleep health in public health agendas across the globe. Lancet Public Health. 2023 Oct;8(10):e820-e826. doi: 10.1016/S2468-2667(23)00182-2. PMID 37777291
- [Derived] Zhang C, Spruyt K, Komolafe M, Mutschelknaus M, DelRosso LM, Steier J. Relationship between shift scheduling, sleep knowledge and sleep quality in medical trainees: protocol for a global cross-sectional survey. J Thorac Dis. 2025 Aug 31;17(8):6339-6347. doi: 10.21037/jtd-2025-291. Epub 2025 Aug 28. PMID 40950851
- See also: Sleep wellbeing (NHS Hospital) — https://www.guysandstthomaseducation.com/project/sleep-looking-after-your-wellbeing
- See also: Working hours (UK Government) — https://www.gov.uk/maximum-weekly-working-hours/print
- See also: The health, safety and wellbeing of shift workers in healthcare environments (NHS) — https://www.nhsemployers.org/system/files/media/Supporting-the-wellbeing-of-shiftworkers-in-healthcare_0.pdf
- See also: Health and Safety Executive: Fatigue (UK Government) — https://www.hse.gov.uk/humanfactors/topics/fatigue.htm
- See also: Tips to consider to fight fatigue at work (Association of Anaesthetists) — https://anaesthetists.org/Fatigue